CLINICAL TRIAL: NCT04648046
Title: Safety and Anti-HIV Activity of Autologous CD4+ and CD8+ T Cells Transduced With a Lentiviral Vector Encoding Bi-specific Anti-gp120 CAR Molecules (LVgp120duoCAR-T) in Anti-retroviral Drug-treated HIV-1 Infection
Brief Title: CAR-T Cells for HIV Infection
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Steven Deeks (Other)
Collaborators: Caring Cross (Unknown)
Responsible Party: Sponsor-Investigator, Steven Deeks, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20-31976
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: HIV Infections
Keywords: HIV; HIV/AIDS; CAR-T cells; HIV cure; HIV reservoir; Immunotherapy
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: The clinical trial is an open-label dose escalating phase I/IIa study of autologous T cells expressing LVgp120duoCAR molecules that target and kill HIV-1 gp120 expressing cells. Participants will be enrolled sequentially in up to three sequentially enrolled cohorts in a 3+3 design. Dose escalation decisions will be made when a minimum of three participants have completed the safety-evaluation period (45 days) at a given dose level. No dose escalation will be allowed in an individual participant, and participants who have dose limiting adverse events will reinstate ART therapy at first available opportunity. There are 3 dose escalation cohorts with the first 3 participants starting at Cohort 1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Dose CAR-T Cells Only (Experimental): Participants will NOT undergo non-ablative conditioning with cyclophosphamide. A single dose of 3 x 10^5 cells/kg LVgp120duoCAR-T cells will be infused. ART will be interrupted immediately after infusion.
  Interventions: Biological: LVgp120duoCAR-T cells, low dose; Other: Analytic Treatment Interruption
- Conditioning + Low Dose CAR-T Cells (Experimental): Participants will undergo non-ablative conditioning with cyclophosphamide. A single dose of 3 x 10^5 cells/kg LVgp120duoCAR-T cells will be infused. ART will be interrupted immediately after infusion.
  Interventions: Drug: Cyclophosphamide; Biological: LVgp120duoCAR-T cells, low dose; Other: Analytic Treatment Interruption
- Conditioning + High Dose CAR-T Cells (Experimental): Participants will undergo non-ablative conditioning with cyclophosphamide. A single dose of 1 x 10^6 cells/kg LVgp120duoCAR-T cells will be infused into the participant. ART will be interrupted immediately after infusion.
  Interventions: Drug: Cyclophosphamide; Biological: LVgp120duoCAR-T cells, high dose; Other: Analytic Treatment Interruption

INTERVENTIONS:
Drug: Cyclophosphamide — Non-ablative conditioning with cyclophosphamide.
  Arms: Conditioning + High Dose CAR-T Cells; Conditioning + Low Dose CAR-T Cells
Biological: LVgp120duoCAR-T cells, low dose — A single dose of 3 x 10^5 cells/kg LVgp120duoCAR-T cells will be infused.
  Arms: Conditioning + Low Dose CAR-T Cells; Low Dose CAR-T Cells Only
Biological: LVgp120duoCAR-T cells, high dose — A single dose of 1 x 10^6 cells/kg LVgp120duoCAR-T cells will be infused.
  Arms: Conditioning + High Dose CAR-T Cells
Other: Analytic Treatment Interruption — HIV antiretroviral therapy medications will be paused.

SUMMARY:
This is a limited-center, open-label dose escalating phase I/IIa study of autologous T cells expressing LVgp120duoCAR molecules in people with HIV infection. It will follow a 3+3 design. Dose escalation decisions will be made when a minimum of three participants have completed the safety-evaluation period (45 days) at a given dose level. Cohort 1 will undergo infusion of a single low-dose regimen of LVgp120duoCAR-T cells. Cohort 2 will undergo non-ablative conditioning with cyclophosphamide, followed by infusion of a single low-dose regimen of LVgp120duoCAR-T cells. Cohort 3 will undergo non-ablative conditioning with cyclophosphamide, followed infusion of a single high-dose regimen of LVgp120duoCAR-T cells. Following administration of the experimental therapy, HIV medications will be paused for participants in each group during an analytic treatment interruption.

DETAILED DESCRIPTION:
A limited-center, open-label dose escalating phase I/IIa study of autologous T cells expressing LVgp120duoCAR molecules will be performed. Participants will be enrolled sequentially in up to three cohorts following a 3+3 design. Dose escalation decisions will be made when a minimum of three participants have completed the safety-evaluation period (45 days) at a given dose level. No dose escalation will be allowed in an individual participant, and participants who have dose limiting adverse events will reinstate ART therapy at first available opportunity.

Following a 3+3 design, each cohort will enroll at least 3 participants. If there are no safety issues with dosing in a cohort, the investigators will proceed to the following cohort. If one participant in a cohort experiences a safety issue, an additional 3 individuals will be enrolled in that cohort to assess safety prior to proceeding to the next cohort. See below for Dose Escalation Procedures.

The first 3 participants start at Cohort 1. Data from Cohort 1 will be submitted for FDA review prior to dosing Cohorts 2 and 3 to determine if cyclophosphamide conditioning is needed.

Cohort 1: Participants will NOT undergo non-ablative conditioning with cyclophosphamide. A single dose of 3 x 105 cells/kg LVgp120duoCAR-T cells will be infused. ART will be interrupted immediately after infusion.

Cohort 2: Participants will undergo non-ablative conditioning with cyclophosphamide. A single dose of 3 x 105 cells/kg LVgp120duoCAR-T cells will be infused. ART will be interrupted immediately after infusion.

Cohort 3: Participants will undergo non-ablative conditioning with cyclophosphamide. A single dose of 1 x 106 cells/kg LVgp120duoCAR-T cells will be infused into the participant. ART will be interrupted immediately after infusion.

Dose Escalation Procedures:

1. If, after 45 days of study treatment, no participant out of the initial 3 in a cohort exhibits a study treatment-related DLT, then the next cohort of participants will be treated at the subsequent cohort.
2. If, after 45 days of study treatment, 1 participant out of the initial 3 in a cohort exhibits a study treatment-related DLT, then up to 3 additional participants will be added at that dose level.
3. If no additional participant develops a study treatment-related DLT (i.e., 1/6 participants with DLT at that dose level), then the next cohort of participants will be treated at the next higher dose level.
4. However, if a second participant develops a study treatment-related DLT, even if it is before there are 6 total participants on that level, then the maximum tolerated dose (MTD) has been exceeded and no additional participants should be added to this or any higher doses. A total of 6 participants should then be treated on the next lowest dose level to ensure its tolerability and to better define the MTD. Thus, the MTD is defined as the highest assigned dose level at which < 2/6 participants have a DLT.
5. If 2 participants in Cohort 1 experience a related DLT, the MTD will have been exceeded and no additional participants will be added at any higher level.
6. If the investigators experience DLTs in Cohort 1, the investigators will de-escalate the dose to 1 x 10^5 cells per kg. If the investigators experience DLTs at the de-escalated dose of 1 x 10^5 cells per kg, the study will stop.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 18 and ≤ 65 years
* HIV-1 infection
* On continuous antiretroviral therapy for at least 12 months without any interruptions of greater than 14 consecutive days, and on a stable regimen that does not include a non-nucleoside reverse transcriptase inhibitor (NNRTI) for at least 4 weeks or any long-acting ART drug that may be active in the participant after ART interruption for up to one year, without plans to modify ART during the study period
* Screening plasma HIV RNA levels below the limit of quantification on all available determinations in past 12 months (isolated single values ≥ 40 but < 200 copies/mL will be allowed if they were preceded and followed by undetectable viral load determinations)
* CD4+ T cell count nadir > 300 cells/mm3
* Screening CD4+ T-cell count ≥ 500 cells/mm3
* Available ART treatment history and the capacity to construct an effective antiretroviral treatment regimen
* Willing to pause ART as part of the study

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
* ART regimen that includes a long-acting anti-HIV drug and/or NNRTI that may be active in the participant for up to one year after ART interruption
* ART regimen that includes protease inhibitor(s) and/or AZT. These drugs may increase the toxicity of cyclophosphamide.
* Any history of an HIV-associated malignancy, including Kaposi's sarcoma and any type of lymphoma, or virus-associated cancers
* History of or current active hepatitis B (HBV) infection defined as positive HBV surface antigen test. A positive anti-HBc regardless of HBsAg status.
* Active hepatitis C (HCV) infection
* Active or latent tuberculosis infection
* Chronic liver disease
* Active and poorly controlled atherosclerotic cardiovascular disease
* Unwillingness to abstain from sex or use barrier protection for any sexual activity during the treatment interruption.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants reporting a new Grade 3 or greater adverse event that is definitely, probably, or possibly related to study treatment within 1 year of product administration. | Within 1 year of product administration
  The primary safety outcome will be the number of participants reporting a new Grade 3 or greater adverse events assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, including signs/symptoms, lab toxicity or clinical event, that is definitely, probably, or possibly related to study treatment within 1 year of product administration.
Number of participants achieving post-treatment control within 36 weeks of product administration. | Week 36
  The primary efficacy outcome will be the proportion of individuals who achieve study-defined post-treatment control. The investigators will define post-treatment control in two ways. First, participants who fail to show any consistent rebound above 400 copies RNA/mL between Weeks 12 and Week 36 will be considered as having achieved post-treatment control. Second, participants who exhibit a rebound and eventually achieve 24 weeks of virus control will be considered as having achieved post-treatment control.

SECONDARY OUTCOMES:
Persistence of LVgp120duoCAR-T cells in blood during therapy | Week 12 through Week 36
  Real-time quantitative polymerase chain reaction (qPCR) will be used to monitor the frequency of circulating CD4+ and CD8+ T cells harboring the integrated LVgp120duoCAR-T gene longitudinally to determine product persistence. This measure will be performed on blood samples.
Persistence of LVgp120duoCAR-T cells in tissues during therapy | Week 12 through Week 36
  Real-time quantitative polymerase chain reaction (qPCR) will be used to monitor the frequency of circulating CD4+ and CD8+ T cells harboring the integrated LVgp120duoCAR-T gene longitudinally to determine product persistence. This measure will be performed on tissue samples collected from volunteers agreeing to lymph node sampling.
Change in quantitative virologic measures of the HIV reservoir pre- and post-therapy | Baseline and 36 weeks
  The HIV reservoir will be measured using methods such as quantitative PCR (qPCR), ultra-sensitive PCR, and/or the intact proviral DNA assay (IPDA) at baseline and time points throughout the study. Changes in the number of copies per 10^6 T cells will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Deeks, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, Davis, Sacramento, California
  - Zuckerberg San Francisco General, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anthony-Gonda K, Ray A, Su H, Wang Y, Xiong Y, Lee D, Block A, Chilunda V, Weiselberg J, Zemelko L, Wang YY, Kleinsorge-Block S, Reese JS, de Lima M, Ochsenbauer C, Kappes JC, Dimitrov DS, Orentas R, Deeks SG, Rutishauser RL, Berman JW, Goldstein H, Dropulic B. In vivo killing of primary HIV-infected cells by peripheral-injected early memory-enriched anti-HIV duoCAR T cells. JCI Insight. 2022 Nov 8;7(21):e161698. doi: 10.1172/jci.insight.161698. PMID 36345941